CLINICAL TRIAL: NCT02907658
Title: A Randomized Efficacy Trial of a Cognitive-Behavioral Intervention to Prevent Internet Use Disorder Onset in Adolescents: the PROTECT Study
Brief Title: Efficacy of Internet Use Disorder Prevention
Acronym: PROTECT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Pädagogische Hochschule Heidelberg (Other)
Collaborators: Dietmar Hopp Stiftung (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PHHD-PROTECT-101030906
Record Dates: First submitted 2016-09-09; First posted 2016-09-20 (Estimated); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: Mental Disorders
Keywords: Internet Use Disorder; Internet Gaming Disorder; Cognitive-Behavioral Intervention; Indicated Prevention; Adolescents; Internet Addiction
MeSH Terms: conditions — Mental Disorders; Internet Addiction Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PROTECT intervention group (Experimental): The PROTECT intervention group receives the preventive intervention PROTECT (4 modules in 4 subsequent weeks à 90 min). Participants are assessed at T1 (baseline), T2 (post treatment, 1-month follow-up), T3 (4-months follow-up), and T4 (12-months follow-up).
  Interventions: Behavioral: PROTECT intervention group
- Assessment-only control group (No Intervention): The assessment-only control group is an observational condition without intervention. Participants are assessed at T1 (baseline), T2 (1-month follow-up), T3 (4-months follow-up), and T4 (12-months follow-up).

INTERVENTIONS:
Behavioral: PROTECT intervention group — The indicated preventive intervention PROTECT consists of a cognitive-behavioral 4-session brief-protocol (90 minutes). It targets empirically identified risk factors of Internet Use Disorder (IUD), i.e. (1) boredom and motivational problems, (2) procrastination and performance anxiety, (3) social behavior and (4) emotion regulation. It addresses both risk-reduction and strength-promotion by cognitive behavioral (CB) interventions such as (1) psychoeducation, (2) cognitive restructuring (identification and modification of dysfunctional cognition), (3) behavior modification (improving problem solving skills, training of functional behavior and reinforcement) as well as (4) improving emotion regulation (training of sensory, imaginative and mindfulness based techniques).
  Arms: PROTECT intervention group

SUMMARY:
Background. The reduction of prevalence rates of Internet Use Disorder (IUD) and its effective treatment are at high priority in both public health and educational policies. School-based preventive interventions facilitate a low-threshold approach for individuals with IUD, who are typically characterized by high therapy avoidance. Moreover, indicated approaches which target adolescents at high-risk show larger effects than universal prevention approaches. Simultaneously, they reduce unnecessary burden for the majority of high-school students that is not at-risk. The PROTECT intervention for indicated prevention of IUD in school settings was developed based on these preventive strategies.

Methods. Three-hundred and forty adolescents, aged 12-18 years, from 40 secondary schools in Germany, screened for high-risk of IUD onset, will be randomly assigned to a) PROTECT intervention group or b) assessment only control group. The tested intervention consists of a cognitive-behavioral 4-session brief-protocol. Follow-up assessments are at 1, 4 and 12 months after admission. Primary outcome is the 12-months incidence rate of IUD. Secondary outcomes are the reduction of IUD and comorbid symptoms and the promotion of problem solving, cognitive restructuring and emotion regulation skills.

Discussion. The indicated preventive intervention PROTECT follows the APA-guidelines for psychological prevention. It is theory- and evidence-based (guideline 1) and addresses both risk-reduction and strength-promotion (guideline 3), it considers current research and epidemiology (guideline 4) and ethical standards (guideline 5) such as professional secrecy and is designed as a systemic intervention (guideline 8) at the school-level. It is expected that the intervention decreases risk of IUD onset (incidence rate).

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 12 to 18 years
* Written informed consent
* High-risk for IUD (Screening: CIUS >= 20)

Exclusion Criteria:

* Current IUD diagnosis or treatment
* Comorbid depression
* Comorbid anxiety disorder (social phobia or performance anxiety)

Ages: 12 Years to 18 Years | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 480 (Actual)
Dates: Start 2015-09; Primary Completion 2018-04 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Internet Use Disorder 12-months incidence rate (Clinical Interview for DSM-5 Diagnosis) | 12 months
  We use a clinical interview (blinded rater) based on the criteria of Internet Gaming Disorder according to the DSM-5 at the 12-month follow-up. We adapted the criteria to assess IUD (including gaming and non-gaming subtypes).
Internet Use Disorder 12-months incidence rate (Self-Report) | 12 months
  We use the German "Computerspielabhängigkeitsskala" (CSAS; Rehbein, Baier, Kleimann & Mößle, 2015), a self-report questionnaire which assesses DSM-5 criteria for Internet Gaming Disorder proposed in DSM-5 section 3 (American Psychiatric Association, 2013): (1) preoccupation, (2) withdrawal, (3) tolerance, (4) unsuccessful attempts to control, (5) loss of interest in other activities, (6) continued excessive use despite problems, (7) deception (8) maladaptive coping, (9) loss of relationship, job, or educational or career opportunities. We adapted the criteria to assess IUD (including gaming and non-gaming subtypes).
Changes in Internet Use Disorder prevalence | baseline, 1 month, 4-months, 12-months
  To measure the IUD prevalence rate over time (at baseline, 1 month, 4-months, 12-months), we use the adapted version of the CSAS questionnaire.

SECONDARY OUTCOMES:
Emotion Regulation | baseline, 1 month, 4-months, 12-months
  For the measurement of emotion regulation the German Questionnaire for Assessment of Emotion Regulation in Children and Adolescents (Fragebogen zur Erhebung der Emotionsregulation bei Kindern und Jugendlichen, FEEL-KJ; Grob & Smolenski, 2011) is used. The questionnaire includes a measure of functional and dysfunctional emotion regulation strategies for the negative emotions fear, sadness and anger.
Depressive Symptoms | baseline, 1 month, 4-months, 12-months
  Depressive symptoms are assessed using the German Depression Inventory for Children and Adolescents (DIKJ; Stiensmeier-Pelster, Braune-Krickau, Schürmann & Duda, 2014; Stiensmeier-Pelster, Schürmann & Duda, 1989). The instrument allows for the detection and estimation of severity of depressive disorders according to the DSM-5 criteria (American Psychiatric Association, 2013).
Comorbid emotional, oppositional, antisocial and attention deficit/ hyperactivity disorders | baseline, 1 month, 4-months, 12-months
  Comorbid Psychopathology is assessed using the Strength and Difficulties Questionnaire (SDQ; Goodman, Meltzer & Bailey, 2003).
  It includes the 5 scales (1) emotional problems, (2) behaviour problems, (3) hyperactivity/ attention deficits, (4) interpersonal problems with peers and (5) prosocial behaviour and can be used for epidemiological research and as an indicator for emotional, oppositional, antisocial and attention deficit/ hyperactivity disorder.
Anxiety Disorders: Social Anxiety | baseline, 1 month, 4-months, 12-months
  We assess social anxiety using the German version of the Social Interaction Anxiety Scale (SIAS; Mattick & Clarke, 1998; Stangier, Heidenreich, Berardi, Golbs & Hoyer, 1999) is used. This questionnaire assesses anxiety in social interactions and al-lows for detection and the estimation of severity of social anxiety disorders.
  2) Performance and school anxiety are assessed with the 7th scale of the German adaption of the Fear Survey Schedule for Children - Revised (Phobiefragebogen für Kinder und Jugendliche, PHOKI Döpfner, Schnabel, Goletz & Ollendick, 2006; Muris & Ollendick, 2002).
Anxiety Disorders: Performance and School Anxiety | baseline, 1 month, 4-months, 12-months
  We assess performance and school anxiety with the 7th scale of the German adaption of the Fear Survey Schedule for Children - Revised (Phobiefragebogen für Kinder und Jugendliche, PHOKI Döpfner, Schnabel, Goletz & Ollendick, 2006; Muris & Ollendick, 2002).
Procrastination | baseline, 1 month, 4-months, 12-months
  Procrastination is assessed with the German Questionnaire for Procrastination (APROF; Höcker, Engberding & Rist, 2013).
Social Behavior and Learning Behavior | baseline, 1 month, 4-months, 12-months
  For ratings of social competent behaviour and academic motivation, we use the German Student Assessment List for Social and Learning Behaviour (SSL; Petermann & Petermann, 2014; Petermann, Petermann & Lohbeck, 2014).
Self-Efficacy | baseline, 1 month, 4-months, 12-months
  Self- efficacy is rated on the German Self-Efficacy Scale (Allgemeine Selbstwirksamkeitserwartung, SWE; Schwarzer & Jerusalem, 1999).

CONTACTS AND LOCATIONS:
Overall Officials: Katajun Lindenberg, PhD, Principal Investigator — University of Education Heidelberg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lindenberg K, Kindt S, Szasz-Janocha C. Effectiveness of Cognitive Behavioral Therapy-Based Intervention in Preventing Gaming Disorder and Unspecified Internet Use Disorder in Adolescents: A Cluster Randomized Clinical Trial. JAMA Netw Open. 2022 Feb 1;5(2):e2148995. doi: 10.1001/jamanetworkopen.2021.48995. PMID 35179587
- [Derived] Wartberg L, Lindenberg K. Predictors of Spontaneous Remission of Problematic Internet Use in Adolescence: A One-Year Follow-Up Study. Int J Environ Res Public Health. 2020 Jan 9;17(2):448. doi: 10.3390/ijerph17020448. PMID 31936677
- [Derived] Lindenberg K, Halasy K, Schoenmaekers S. A randomized efficacy trial of a cognitive-behavioral group intervention to prevent Internet Use Disorder onset in adolescents: The PROTECT study protocol. Contemp Clin Trials Commun. 2017 Mar 29;6:64-71. doi: 10.1016/j.conctc.2017.02.011. eCollection 2017 Jun. PMID 29740637
- [Derived] Lindenberg K, Halasy K, Szasz-Janocha C, Wartberg L. A Phenotype Classification of Internet Use Disorder in a Large-Scale High-School Study. Int J Environ Res Public Health. 2018 Apr 12;15(4):733. doi: 10.3390/ijerph15040733. PMID 29649137